CLINICAL TRIAL: NCT06237010
Title: Impact of Covid-19 on Occupational Dermato-allergology Consultations of Health Peronnel
Acronym: ÉPIDERMAPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ÉPIDERMAPS-COVID-19
Record Dates: First submitted 2024-01-31; First posted 2024-02-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Dermatoses; Health Workers
Keywords: COVID-19; Dermatoses; Contact dermatitis; Occupational dermatitis
MeSH Terms: conditions — Skin Diseases; COVID-19; Dermatitis, Contact; Dermatitis, Occupational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Occupational dermatitis is the second most common occupational disease in Europe, with a notable prevalence among healthcare workers-approximately 20% of whom are affected. However, these figures may be underestimated due to underreporting. Despite the presumed scale of the problem, there is no recent European data providing real numbers. This study seeks to address the knowledge gap regarding the impact of the COVID-19 pandemic on occupational dermatitis within the healthcare workers population.

EPIDERMAPS is a retrospective cohort study that analyzes data from two specialized centers in the Paris region. The primary goal is to assess changes in the proportion of dermatology-allergology consultations among healthcare workers before and after the COVID-19 pandemic. Secondary objectives include evaluating the pandemic's effect on occupational dermatoses incidences, attributed to increased PPE and hygiene products usage. The major focus will be on work-related allergic contact dermatitis, irritant contact dermatitis, contact urticaria, acne, and rosacea. The latter objective is to identify new allergens or contributing factors.

Participants include active healthcare workers aged 18 or older who sought consultations for dermatological or dermatology-allergology related motifs between March 15, 2017, and March 15, 2023. Exclusions apply for patients who have consulted for other than dermatology-allergology related motif and those opposing to participate. Data will be stored, anonymized, and analyzed using EasyMedStat. Data collection is scheduled between March and December 2024.

This research aims to offer insights into COVID-19's dermatologic and allergic effects on healthcare professionals, informing future preventive measures and enhanced care strategies.

DETAILED DESCRIPTION:
Occupational dermatoses include several dermatological conditions, the most common are allergic contact dermatitis, irritant contact dermatitis, contact urticaria, acne, and rosacea. Occupational dermatitis is the second most common occupational disease in Europe, with a notable prevalence among healthcare workers-approximately 20% of whom are affected. However, these figures may be underestimated due to underreporting. Despite the presumed scale of the problem, there is no recent European data providing real numbers. This study seeks to address the knowledge gap regarding the impact of the COVID-19 pandemic on occupational dermatitis within the healthcare workers population.

EPIDERMAPS is a retrospective cohort study that analyzes data from two Parisian centers specialized in occupational dermatology and allergology - Centre Hospitalier Intercommunal de Créteil and l'Hôpital Hôtel Dieu in Paris. Both centers are recognized at the national level as the Occupational and Environmental Disease Consultation Center (Centre de Consultation de Pathologies Professionnelles et de l'Environnement).

The primary goal is to analyze the impact of the COVID-19 on the proportion of dermatology-allergology consultations of healthcare workers in relation to the total number of consultations in these two centers, before and after the pandemic.

Secondary objectives include:

* Analysis of the impact of COVID-19 on the incidence of dermatoses induced by the increased use of surgical masks and gloves, increased handwashing, and the heightened use of hydro-alcoholic solutions and surface disinfectants among healthcare personnel. The major focus will be on allergic contact dermatitis, irritant contact dermatitis, contact urticaria, acne and rosacea.
* Analysis of the impact of COVID-19 on the contact allergic sensitization to components of surgical masks, gloves, soaps, disinfectant cleansers, and hydroalcoholic solutions among healthcare personnel.
* Identification of new allergens or new factors causing dermatoses among healthcare personnel following the COVID-19 epidemic.

The Inclusion criteria require to be an active healthcare worker aged 18 or older at the date of the first consultation. Further criteria are to have consulted for dermatological or dermatology-allergology related motifs between March 15, 2017, and March 15, 2023. Exclusions apply for non-healthcare workers, patients who have consulted for other than dermatology-allergology related motif, and those opposing to participate. Patient identification involves querying the National Network for Surveillance and Prevention of Occupational Diseases (RNV3P, Réseau National de Vigilance et de Prévention des Pathologies professionnelles). Eligible patients will be informed by mail, and if no opposition expressed, their data will be collected and stored anonymously for analysis. Patient data will be collected from medical records, anonymized, and stored securely. Data collection is programmed from March to December 2024. The study comprises 471 patients from two centers.

The collected data will include:

* Age at the first consultation
* Date of the first consultation
* Date of birth (month and year)
* Gender
* Occupation
* Duration in the profession
* Diagnosed condition(s)
* Date of symptom onset
* Nature of symptoms
* Location of lesions
* Identified aggravating/triggering factors
* Professional rhythm of lesions
* History, such as:

  * Atopic dermatitis
  * Asthma
  * Rhinoconjunctivitis
  * Contact dermatitis
  * Documented allergic sensitization to an allergen
  * Urticaria
  * Acne
  * Rosacea
* Patch test results and their relevance
* Prick test results
* Socio-professional outcome (job accommodation, job change, career reorientation, etc.)

Statistical analyses will use EasyMedStat to respond to the primary and secondary objectives.

The study has been officially approved by the Local Ethics Committee (CEL) of Créteil on the December 19th, 2023.

In conclusion, this research aims to provide new data on COVID-19's dermatologic and allergic effects on healthcare professionals, informing future preventive measures and enhanced care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consulted for the first time between 15th march 2017 and 15th march 2023 for an occupational dermato-allergological problem ;
* Active subjects and occupying a health personnel position defined according to the Public Health Code ;
* Over 18 years old at the first consultation, with no upper limit
* Having not expressed their opposition to participate in the study.

Exclusion Criteria:

* Patients who consulted for an other problem than occupational dermato-allergological problem ;
* Patients who not consulted for the first time between 15th march 2017 and 15th march 2023.
* Patients without occupational activity the day of the first consultation
* Patients who opposite to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consulted for the first time between 15th march 2017 and 15th march 2023 for an occupational dermato-allergological problem and occupying a health personnel position.
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Proportion of occupational dermato-allergology consultations | Day 1
  Proportion of occupational dermato-allergology consultations

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Hôtel Dieu, Paris

IPD SHARING:
Plan to Share IPD: No